CLINICAL TRIAL: NCT02964039
Title: A Novel Mechanics-based Intervention to Improve Post-stroke Gait Stability
Brief Title: A Novel Mechanics-based Intervention to Improve Post-stroke Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N2256-R; RX002256 (Other Grant/Funding Number: VA ORD)
Record Dates: First submitted 2016-11-04; First posted 2016-11-15 (Estimated); Results first posted 2021-07-28 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-12

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Error reduction (Experimental): Participants will complete a 12-week training program, in which they practice walking on a treadmill for 30-minutes during twice-weekly training sessions. During these sessions, participants will interface with a custom-built force-field able to exert mediolateral forces on the legs, which will be in "error reduction" mode. This training period will be followed by a 12-week follow-up period. Five assessment sessions will be interspersed throughout this total 24-week period.
  Interventions: Behavioral: Error reduction
- Error augmentation (Experimental): Participants will complete a 12-week training program, in which they practice walking on a treadmill for 30-minutes during twice-weekly training sessions. During these sessions, participants will interface with a custom-built force-field able to exert mediolateral forces on the legs, which will be in "error augmentation" mode. This training period will be followed by a 12-week follow-up period. Five assessment sessions will be interspersed throughout this total 24-week period.
  Interventions: Behavioral: Error augmentation
- Activity matched control (Sham Comparator): Participants will complete a 12-week training program, in which they practice walking on a treadmill for 30-minutes during twice-weekly training sessions. During these sessions, participants will interface with a custom-built force-field able to exert mediolateral forces on the legs, which will be in "transparent" mode. This training period will be followed by a 12-week follow-up period. Five assessment sessions will be interspersed throughout this total 24-week period.
  Interventions: Behavioral: Activity matched control

INTERVENTIONS:
Behavioral: Error reduction — During training sessions, a custom-built force-field will exert forces on the legs while participants walk. These forces will push the legs toward mechanically-appropriate mediolateral locations, having the effect of reducing the errors in foot placement that are often present among individuals who have experienced a stroke.
  Arms: Error reduction
Behavioral: Error augmentation — During training sessions, a custom-built force-field will exert forces on the legs while participants walk. These forces will push the legs away from mechanically-appropriate mediolateral locations, having the effect of amplifying the errors in foot placement that are often present among individuals who have experienced a stroke.
  Arms: Error augmentation
Behavioral: Activity matched control — During training sessions, participants will interface with a custom-built force-field while they walk. The force-field will essentially get out of the way, producing minimal forces on the legs, and having no direct effect on the errors in foot placement that are often present among individuals who have experienced a stroke.
  Arms: Activity matched control

SUMMARY:
The purpose of this study is to determine whether a novel treadmill training intervention can improve the gait stabilization strategy used by individuals who have experienced a stroke.

DETAILED DESCRIPTION:
Every year, approximately 15,000 American Veterans experience a stroke, with an estimated cost of acute and follow-up care in the hundreds of millions of dollars. Following a stroke, the restoration or improvement of walking is a high-ranking goal among patients, but only about half of the population is able to return to typical levels of community ambulation. The resultant decrease in independent mobility is strongly associated with a decline in quality of life. Gait instability is a common contributor to limited mobility through either an increased fall-risk or fear of falling, but current interventions to address post-stroke gait instability have had limited success. This project will conduct initial testing of a novel elastic force-field designed to improve post-stroke gait stability through targeted motor learning. The results of these experiments will serve as the basis for the development of novel gait rehabilitation techniques, which have the potential to increase the quality of life of thousands of Veterans and save millions of dollars.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Experience of a stroke 6 months prior to participation
* Preferred overground gait speed of at least 0.2 m/s
* Ability to walk at self-selected speed for 3 minutes without a cane or walker
* Provision of informed consent.

Exclusion Criteria:

* Resting heart rate above 110 beats/min
* Resting blood pressure higher than 200/110 mm Hg
* History of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living
* Preexisting neurological disorders or dementia
* History of major head trauma
* Legal blindness or severe visual impairment
* Life expectancy <1 yr; 8)
* History of deep vein thrombosis or pulmonary embolism within 6 months
* Uncontrolled diabetes with recent weight loss, diabetic coma, or frequent insulin reactions
* Orthopedic injuries or conditions (e.g. joint replacements) in the lower extremities with the potential to alter the gait pattern.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C. Dean, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified, anonymized data sets will be available to other investigators or members of the public upon request. These data sets will be made available upon completion of data collection, processing, and initial statistical analyses. The data sets will include physiological measures related to functional mobility, as well as the results of clinical tests.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and enrolled between February 2017 and October 2019 from a database housed at the Medical University of South Carolina. Individuals in this database had previously experienced a stroke, and had agreed to be contacted for participation in research studies.
Pre-assignment Details: Of the 93 participants who were assessed for eligibility, 54 met the study's inclusion criteria and were interested in participating in the intervention. These 54 participants were randomized to one of the three study arms.
Period: Overall Study
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Started | 18 | 18 | 18
Received Allocated Intervention | 15 | 17 | 14
Completed (Re-assessed after 12-week follow-up period) | 14 | 17 | 13
Not Completed | 4 | 1 | 5
Not completed — Medical reason unrelated to study participation | 1 | 0 | 3
Not completed — Research shutdown due to pandemic | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (13) | 57 (13) | 57 (14) | 59 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 9 | 24
  Male | 9 | 12 | 9 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 18 | 18 | 18 | 54
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 8 | 21
  White | 12 | 10 | 10 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Affected leg [Count of Participants; unit: Participants]
  Left leg | 10 | 9 | 10 | 29
  Right leg | 8 | 9 | 8 | 25
Time since stroke [Mean (Standard Deviation); unit: months] — The number of months since the participant experienced a stroke at the time of study enrollment, based on information stored in the participant database used for recruitment
  months | 53 (48) | 53 (46) | 56 (57) | 54 (50)
Height [Mean (Standard Deviation); unit: inches] | 66 (4) | 68 (4) | 67 (4) | 67 (4)
Weight [Mean (Standard Deviation); unit: pounds] | 187 (49) | 189 (44) | 181 (39) | 186 (43)
Partial Correlation Between Pelvis Displacement and Paretic Step Width During Gait [Mean (Standard Deviation); unit: Correlation Coefficient] — This measure relates the mechanical state of the body at the start of each step (mediolateral pelvis displacement and velocity of the pelvis relative to the stance foot) to the step width at the end of the step. Specifically, the partial linear correlation between pelvis displacement and step width was calculated, accounting for variation in pelvis velocity. Population: Here, we present the baseline measures for only those participants who completed the intervention.
  Correlation Coefficient
    number analyzed (Participants) | 14 | 17 | 13 | 44
    (all) | 0.44 (0.10) | 0.34 (0.19) | 0.51 (0.10) | 0.43 (0.16)
Functional Gait Assessment [Mean (Standard Deviation); unit: Score on a scale] — The Functional Gait Assessment is a standardized clinical test used to assess balance during a variety of walking tasks. Possible scores range from 0 to 30, with 30 representing the best balance performance. The total possible score of 30 represents the sum of 10 possible subscores for each walking task, with each having a possible range from 0 to 3. Population: Here, we present the baseline measures for only those participants who completed the intervention.
  Score on a scale
    number analyzed (Participants) | 14 | 17 | 13 | 44
    (all) | 15.5 (3.2) | 13.8 (5.2) | 13.5 (5.0) | 14.3 (4.6)
Activities-specific Balance Confidence scale [Mean (Standard Deviation); unit: Score on a scale] — This measure is a common clinical assessment of balance self-efficacy during a variety of movement tasks that participants may experience in the community. Possible scores range from 0 to 100, with 100 representing the best self-efficacy. Scores are calculated as the mean of 16 subscores, each of which ranges from 0 to 100 and represents self-efficacy during a different movement task. Population: Here, we present the baseline measures for only those participants who completed the intervention.
  Score on a scale
    number analyzed (Participants) | 14 | 17 | 13 | 44
    (all) | 65.7 (22.2) | 69.8 (12.4) | 69.3 (15.3) | 68.3 (16.6)
Walking speed (10-meter walk test) [Mean (Standard Deviation); unit: meters per second] — Population: Here, we present the baseline measures for only those participants who completed the intervention.
  meters per second
    number analyzed (Participants) | 14 | 17 | 13 | 44
    (all) | 0.84 (0.21) | 0.73 (0.31) | 0.78 (0.31) | 0.78 (0.28)
Fall incidence (self reported over previous year) [Count of Participants; unit: Participants] — Population: Here, we present the baseline measures for only those participants who completed the intervention.
  Participants
    number analyzed (Participants) | 14 | 17 | 13 | 44
    (all) | 6 | 7 | 7 | 20
Fear of falling (self-reported) [Count of Participants; unit: Participants] — Population: Here, we present the baseline measures for only those participants who completed the intervention.
  Participants
    number analyzed (Participants) | 14 | 17 | 13 | 44
    (all) | 5 | 7 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Partial Correlation Between Pelvis Displacement and Paretic Step Width During Gait (Change From Baseline)
Description: A custom measure that quantifies the strength of the relationship between body mechanics and foot placement. This measure falls within a relatively narrow range among neurologically intact controls, but is substantially reduced in some individuals who have experienced a stroke, indicating a reduced ability to stabilize their gait pattern. This measure relates the mechanical state of the body at the start of each step (mediolateral pelvis displacement and velocity of the pelvis relative to the stance foot) to the step width at the end of the step. Specifically, the partial linear correlation between pelvis displacement and step width was calculated, accounting for variation in pelvis velocity.
  The change in this measure relative to baseline is calculated at four time points (after 4, 8, 12, and 24 weeks).
Time Frame: baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks
Population: The total of 44 participants analyzed corresponds to the participants who completed the intervention and follow-up assessment.
Measure: Mean (Standard Deviation); unit: Correlation coefficient
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Number analyzed (Participants) | 14 | 17 | 13
Correlation coefficient
  4-week assessment | -0.02 (0.22) | 0.12 (0.20) | -0.04 (0.14)
  8-week assessment | 0.05 (0.15) | 0.11 (0.20) | -0.02 (0.16)
  12-week assessment | 0 (0.08) | 0.08 (0.18) | 0.01 (0.12)
  Follow-up assessment (after 12 weeks) | -0.01 (0.16) | 0.11 (0.18) | 0 (0.14)
Statistical Analysis 1: Comparison: Error Reduction vs Error Augmentation vs Activity Matched Control; Test type: Superiority; p = 0.047, ANOVA — A priori threshold: 0.05; 0.047 is the main effect of group from a 2-way ANOVA that also included time (p=0.77) as a within-subjects factor

2. Secondary Outcome: Functional Gait Assessment (Change From Baseline)
Description: A commonly-used clinical test to quantify balance and stability during various walking tasks. The minimum value is 0, the maximum value is 30, and higher scores indicate better outcomes. The total maximum value of 30 is calculated as the sum of 10 subscores, each of which has a scoring range of 0-3 and represents a distinct walking task.
  The change in this measure relative to baseline is calculated at four time points (after 4, 8, 12, and 24 weeks).
Time Frame: baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Number analyzed (Participants) | 14 | 17 | 13
score on a scale
  4-week assessment | 0.1 (1.8) | 1.5 (2.3) | 1.6 (2.1)
  8-week assessment | 0.8 (2.3) | 1.9 (2.7) | 2.5 (2.8)
  12-week assessment | 1.5 (2.5) | 2.9 (1.9) | 2.1 (1.8)
  Follow-up assessment (after 12 weeks) | 1.0 (2.5) | 2.2 (2.5) | 1.9 (3.5)
Statistical Analysis 1: Comparison: Error Reduction vs Error Augmentation vs Activity Matched Control; Test type: Superiority; p = 0.16, ANOVA — A priori threshold: 0.05; 0.16 is the main effect of group from a 2-way ANOVA that also included time (p=0.023) as a within-subjects factor

3. Secondary Outcome: Activities-specific Balance Confidence Scale (Change From Baseline)
Description: A commonly-used clinical scale that quantifies an individual's confidence in performing various tasks requiring balance. The minimum value is 0, the maximum value is 100, and higher scores indicate a better outcome. The overall score is calculated as the mean of 16 subscores, each of which can range of 0 to 100 and represents self-efficacy at a distinct movement task.
  The change in this measure relative to baseline is calculated at four time points (after 4, 8, 12, and 24 weeks).
Time Frame: baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Number analyzed (Participants) | 14 | 17 | 13
score on a scale
  4-week assessment | 2.2 (11.2) | -0.6 (6.9) | 3.7 (10.3)
  8-week assessment | 2.5 (12.9) | -1.2 (4.9) | 4.1 (16.2)
  12-week assessment | 6.1 (16.4) | 2.8 (6.8) | 5.4 (12.5)
  Follow-up assessment (after 12 weeks) | 8.1 (14.7) | 4.6 (7.9) | 3.7 (22.8)
Statistical Analysis 1: Comparison: Error Reduction vs Error Augmentation vs Activity Matched Control; Test type: Superiority; p = 0.64, ANOVA — A priori threshold: 0.05; 0.64 is the main effect of group from a 2-way ANOVA that also included time (p=0.024) as a within-subjects factor

4. Secondary Outcome: 10-meter Walk Test (Change From Baseline)
Description: A commonly-used clinical test to quantify general gait function. Walking speed is measured during the middle 6-meter portion of a 10-meter straight line path.
  The change in this measure relative to baseline is calculated at four time points (after 4, 8, 12, and 24 weeks).
Time Frame: baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Number analyzed (Participants) | 14 | 17 | 13
meters per second
  4-week assessment | 0.01 (0.08) | 0.03 (0.08) | 0.03 (0.08)
  8-week assessment | 0.02 (0.10) | 0.04 (0.07) | 0.04 (0.10)
  12-week assessment | 0.05 (0.14) | 0.02 (0.08) | 0.06 (0.10)
  Follow-up assessment (after 12 weeks | 0.01 (0.15) | 0.01 (0.11) | 0.01 (0.11)
Statistical Analysis 1: Comparison: Error Reduction vs Error Augmentation vs Activity Matched Control; Test type: Superiority; p = 0.92, ANOVA — A priori threshold: 0.92; 0.92 is the main effect of group from a 2-way ANOVA that also included time (p=0.076) as a within-subjects factor

5. Secondary Outcome: Fall Incidence
Description: Self-report history of fall occurrence, quantified by the average number of falls per participant in each group during the 12-week period that followed completion of the study's intervention component
Time Frame: 6 months (during 12 week follow-up period)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Falls per participant
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Number analyzed (Participants) | 14 | 17 | 13
Falls per participant | 0.50 (0.20) | 0.29 (0.14) | 0.62 (0.23)
Statistical Analysis 1: Comparison: Error Reduction vs Error Augmentation vs Activity Matched Control; Test type: Superiority; p >= 0.22, Mixed Models Analysis — A priori threshold: 0.05; We compared incident rates assuming a negative binomial distribution with leas squares means estimates predicted via generalized linear model

6. Secondary Outcome: Fear of Falling
Description: Self-report statement of whether a participant has a fear of falling
Time Frame: 6 months (at completion of 12-week Follow-up period)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
Number analyzed (Participants) | 14 | 17 | 13
Participants | 4 | 5 | 4
Statistical Analysis 1: Comparison: Error Reduction vs Error Augmentation vs Activity Matched Control; Test type: Superiority; p = 0.99, Chi-squared — A priori threshold: 0.05

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a three-year period, corresponding from the time when the first participant was enrolled into the intervention to the time when the overall intervention ended.
Description: We adhered to guidance provided by the Medical University of South Carolina Institutional Review Board; in order for an event to be classified as a reportable adverse event, it cannot be "the expected natural progression of any underlying disease, disorder, or condition of the subject experiencing the adverse event and the subject's predisposing risk factor profile for the adverse event". While we tracked falls, they are thus not included as adverse events.
Arm/Group | Error Reduction | Error Augmentation | Activity Matched Control
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 1/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Error Reduction (N=18) | Error Augmentation (N=18) | Activity Matched Control (N=18)
Stroke (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — A participant was diagnosed with an acute ischemic stroke in the left middle cerebral artery while enrolled in the study. No major deficits resulted following the stroke. The participant was withdrawn from the study.

LIMITATIONS AND CAVEATS:
The overall dropout rate of this study was increased by the research shutdown with the coronavirus pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/39/NCT02964039/Prot_SAP_000.pdf